CLINICAL TRIAL: NCT03139071
Title: Coffee Consumption and Coronary Artery Calcium Score: Results From the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil)
Brief Title: Coffee Consumption and Coronary Artery Calcium Score
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Dirce Maria Lobo Marchioni, Professor, University of Sao Paulo
Other Study IDs: marchioni2017
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Atherosclerosis; Cardiovascular Diseases
Keywords: coffee consumption; cardiovascular diseases; coronary artery calcium; subclinical atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Coffee is one of the dietary factors associated with cardiovascular disease (CVD) but its role in the cardiovascular system is not yet clear. Moreover, available evidence for the relation between coffee intake with subclinical atherosclerosis is limited and inconsistent. The aim of this study was to evaluate the association between habitual coffee consumption and the presence of subclinical atherosclerosis measured as coronary artery calcium (CAC) in the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil). This is a cross-sectional study based on baseline data from participants of the cohort ELSA-Brasil. In this analysis, only participants living in São Paulo with no prior history of CVD aged 35 to 74 years who underwent a CAC measurement (n=4,426) were included. Dietary data were collected using a validated food frequency questionnaire. Coronary calcification was detected with computed tomographic and it was expressed as Agatston units. CAC was further categorized as 0 or >0, and <100 or ≥100.

DETAILED DESCRIPTION:
The Longitudinal Study of Adult Health (ELSA-Brasil) is a cohort study designed to identify risk factors for diabetes and CVD. Briefly, the cohort comprises 15,105 civil servants, aged 35 to 74 years at baseline, who were sampled from universities or research institutions located in six cities (Belo Horizonte, Porto Alegre, Rio de Janeiro, Salvador, São Paulo, and Vitoria) of three different regions of Brazil. Baseline assessment was conducted from August 2008 to December 2010 and consisted of an approximately 7-hour evaluation, which included personal interviews conducted by trained personnel. These interviews focused on sociodemographic characteristics, health and medical history, occupational exposure, family history of disease, reproductive health, health care, psychosocial factors, body weight history and body image, food consumption, smoking, alcohol consumption, physical activity, medication use, cognitive function, mental health, and clinical and laboratory measurements. In addition, the participants at the ELSA-Brasil site in São Paulo were invited to perform a computed tomographic (CT) examination to quantify coronary artery calcium (CAC).

Thus, for the current investigation, only participants of the ELSA-Brasil of São Paulo Research Center who submitted to CAC determination (n=4,549) were included. In addition, in the present analysis, we considered individuals without missing data at baseline for coffee intake, and no self-reported history of cardiovascular disease defined as prior myocardial infarction, angina, stroke, heart failure, and coronary revascularization. Therefore, the final study sample comprised 4,426 individuals who submitted to CAC measurements and did not fulfill exclusion criteria to participate in this subset of the study.

The ELSA-Brasil protocol was approved at all six centers by the institutional review boards addressing research in human participants. All the subjects signed a written informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* For the current investigation, only participants of the ELSA-Brasil of São Paulo Research Center who submitted to CAC determination (n=4,549) were included.

Exclusion Criteria:

* Missing data at baseline for coffee intake, and self-reported history of cardiovascular disease defined as prior myocardial infarction, angina, stroke, heart failure, and coronary revascularization.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Longitudinal Study of Adult Health (ELSA-Brasil) is a cohort study that comprises 15,105 civil servants, aged 35 to 74 years at baseline, who were sampled from universities or research institutions located in six cities (Belo Horizonte, Porto Alegre, Rio de Janeiro, Salvador, São Paulo, and Vitoria) of three different regions of Brazil.
  The participants at the ELSA-Brasil site in São Paulo were invited to perform a computed tomographic (CT) examination to quantify coronary artery calcium (CAC).
  Thus, for the current investigation, only participants of the ELSA-Brasil of São Paulo Research Center who submitted to CAC determination (n=4,549) were included. Therefore, the final study sample comprised 4,426 individuals who submitted to CAC measurements and did not fulfill exclusion criteria to participate in this subset of the study.
Sampling Method: Non-Probability Sample
Enrollment: 4426 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
subclinical atherosclerosis | Through study completion, an average of 2 to 4 years.
  The presence and severity of subclinical atherosclerosis were measured as coronary artery calcium. The ELSA-Brasil participants from the São Paulo site underwent noncontrast computed tomographic (CT) for CAC score evaluation. The scans were performed using a 64 detector CT scanner (Brilliance 64; Philips Healthcare, Philips Healthcare, Best, Netherlands). The measurement of the CAC score was calculated using a threshold of 130 HU and expressed in Agatston units.

CONTACTS AND LOCATIONS:
Locations (1):
- Dirce Maria Marchioni, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No